CLINICAL TRIAL: NCT01872936
Title: Phase 2, Open-Label, Clinical Trial of Miravirsen Sodium in Combination With Telaprevir and Ribavirin in Null Responders to Pegylated-Interferon Alpha Plus Ribavirin Subjects With Chronic Hepatitis C Virus Genotype 1 Infection
Brief Title: Miravirsen in Combination With Telaprevir and Ribavirin in Null Responder to Pegylated-Interferon Alpha Plus Ribavirin Subjects With Chronic Hepatitis C Virus Infection
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Santaris Pharma A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SPC3649-205
Record Dates: First submitted 2013-06-03; First posted 2013-06-07 (Estimated); Last update posted 2014-11-18 (Estimated); Status verified 2014-11

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — miravirsen; telaprevir; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Miravirsen every other week dosing (Other): Miravirsen will be dosed as single subcutaneous injections. Subjects will receive 5 weekly doses at 7 mg/kg, then 6 every other week doses at 5 mg/kg in combination with telaprevir and ribavirin.
  Interventions: Drug: Miravirsen; Drug: Telaprevir; Drug: Ribavirin
- Miravirsen monthly dosing (Other): Miravirsen will be dosed as single subcutaneous injections. Subjects will receive 5 weekly doses at 7 mg/kg, then 3 monthly doses at 7 mg/kg in combination with telaprevir and ribavirin.
  Interventions: Drug: Miravirsen; Drug: Telaprevir; Drug: Ribavirin

INTERVENTIONS:
Drug: Miravirsen
  Other Names: SPC3649; Miravirsen sodium
Drug: Telaprevir
  Other Names: Incivek
Drug: Ribavirin
  Other Names: Copegus

SUMMARY:
The purpose of this open-label study is to assess the safety, tolerability, antiviral activity, genotype resistance associated with virological failure, pharmacokinetics and pharmacodynamics of two dose regimens of miravirsen in combination with telaprevir and ribavirin in subjects with hepatitis C virus genotype 1 infection who are null responder to pegylated-interferon alpha and ribavirin.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic hepatitis C genotype 1 infection
* BMI 18 and 38 kg/m2
* Null responder to pegylated interferon alpha and ribavirin

Exclusion Criteria:

* Co-infection with hepatitis B virus (HBV) or human immunodeficiency virus (HIV)
* Significant liver disease in addition to hepatitis C
* Decompensated liver disease medical history or current clinical features
* Histologic evidence of hepatic cirrhosis
* Concurrent clinically significant medical diagnosis (other than CHC)
* Concurrent social conditions (e.g. drugs of abuse, alcohol excess, poor living accommodation)
* Clinically significant illness within 30 days preceding entry into the study
* Participated in an investigational drug study within 30 days or 5 half-lives, whichever is longer, prior to the start of study medication
* History of clinically significant allergic drug reactions

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2013-06; Primary Completion 2015-01 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
The proportion of subjects with a Sustained Virological Response at 24 weeks after the end of therapy. | 42 weeks

SECONDARY OUTCOMES:
The proportion of subjects with undetectable HCV RNA levels at end of treatment. | 18 weeks
The proportion of subjects with a Sustained Virological Response at 12 and 48 weeks after the end of therapy. | 66 Weeks
Change in HCV RNA levels from baseline throughout the study. | 66 Weeks
The proportion of subjects who experience virological failure throughout the study. | 66 Weeks

OTHER OUTCOMES:
Viral resistance analysis at baseline and throughout the study. | 66 Weeks
  The miR-122 seed sites in HCV RNA from subjects at baseline and following viral breakthrough or relapse will be subjected to genotypic sequence analysis.
Plasma pharmacokinetics (AUC, Cmax, tmax) for miravirsen, telaprevir, and ribavirin levels will be determined. | 31 Weeks
  A single sample will be collected at select study visits for all subjects through Week 31. A subset of subjects will participate in extended PK sampling for up to 5 hours at select study visits and for up to 24 hours after the last dose of miravirsen.
Urine pharmacokinetics for miravirsen levels will be determined. | Up to 16 Weeks
  Urine pharmacokinetics (AUC, Cmax, tmax) for miravirsen levels will be measured in a subset of subjects for up to 24 hours after the last dose of miravirsen.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Hodges, MD, Study Director — Santaris Pharma A/S
Locations (3):
- United States (2):
  - The Liver Institute at Methodist Dallas Medical Center, Dallas, Texas
  - Research Specialists of Texas, Houston, Texas
- Fundacion de Investigacion de Diego, San Juan, Puerto Rico